CLINICAL TRIAL: NCT02884804
Title: Study of Biological Determinants of Bleeding Postpartum : Predictive Role in the Number of Immature Platelets
Brief Title: Study of Biological Determinants of Bleeding Postpartum
Acronym: HPP-IPF
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: HPP-IPF (RB 11.080)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum Hemorrhage; Immature platelet
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PLASMA
Oversight: Data Monitoring Committee: No

SUMMARY:
At the entry of the delivery room, a standard blood analysis will be performed (Blood count, PT, aPTT, Fibrinogen, and D-Dimer) for each women (if they are agree), according to the center's practices.

The percentage of the immature platelets is a an additional parameter on the hemogram.

The clinical assessments (recorded in medical records) and biological values will be used to determine if there is a correlation between these data and the occurrence of postpartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Woman giving birth in a maternity of Finistère

Exclusion Criteria:

* Refuse to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Woman giving birth in a maternity of Finistère (France)
Sampling Method: Non-Probability Sample
Enrollment: 3599 (Actual)
Dates: Start 2011-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Postpartum Hemorrhage | Volume of blood loss up to 24 hours after delivery and / or weight compresses collected at delivery, and / or diagnosis of the clinician
Percentage of immature platelets | Percentage of immature platelets just before the entry in the birth room

CONTACTS AND LOCATIONS:
Overall Officials: PAN-PETESCH Brigitte, Dr., Principal Investigator — CHRU de BREST
Locations (1):
- CHRU de BREST, Brest, France